CLINICAL TRIAL: NCT06401187
Title: Evaluation of Patient Satisfaction and Maximum Biting Force of Three Different Constructed Bars in Implant Overdenture in One Year Follow-up
Brief Title: Patient Satisfaction and Maximum Biting Force in Co-Cr Bar Implant Overdenture
Acronym: bar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, mona nabawy, lecturer assistant, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 644; Amr Esmail (Other: minia university); shaimaa Radwan (Other: Minia UNiversity)
Record Dates: First submitted 2024-04-30; First posted 2024-05-06 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Dental
Keywords: implants,; Milled; 3D printed; Patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Co-Cr conventional technique cast bar attachments (Active Comparator): conventional technique cast bar attachments
  Interventions: Other: Bar overdenture
- Co-Cr CAD/CAM milled bar attachments (Experimental): Co-Cr CAD/CAM milled bar attachments
  Interventions: Other: Bar overdenture
- Co-Cr CAD/CAM 3D bar attachments (Experimental): Co-Cr CAD/CAM 3D bar attachments
  Interventions: Other: Bar overdenture

INTERVENTIONS:
Other: Bar overdenture — use of bar attachments as retentive mean of denture
  Other Names: bar overdenture implants

SUMMARY:
Statement of problem. Patient satisfaction and maximum biting force from patients who wear 2-implant-retained overdentures with different constructed bar attachments can be improved.

Purpose. This randomised controlled clinical trial assessed patient satisfaction and maximum biting force with three differently constructed bar-retained overdentures (conventional casting, Milling and 3D printing CAD/CAM techniques) within a one-year follow-up.

Material and methods. A total of 60 implants were placed in 30 mandibular jaws(30 participants). The jaws were randomly assigned to 1 of the 3 treatment groups: a 10 conventional technique cast Co-Cr bar attachment, a 10 Co-Cr CAD/CAM milled bar attachment, and a 10 Co-Cr CAD/CAM 3D-printed bar attachment all groups were connected to 2 implants in the canine area. Patient satisfaction was tested after 6 months, and 12 months for each group; the results were collected, tabulated, and statistically analysed using a Pair-wise comparisons test and the Kruskal-Wallis test. Maximum biting force was tested at baseline,3 months, 6 months, and 12 months for each group; the results were collected, tabulated, and statistically analysed using a Pair-wise comparisons test and ANOVA test.

DETAILED DESCRIPTION:
A total of 60 implants were placed in 30 mandibular jaws(30 participants). The jaws were randomly assigned to 1 of the 3 treatment groups: a 10 conventional technique cast Co-Cr bar attachment, a 10 Co-Cr CAD/CAM milled bar attachment, and a 10 Co-Cr CAD/CAM 3D-printed bar attachment all groups were connected to 2 implants in the canine area. Patient satisfaction was tested after 6 months, and 12 months for each group; the results were collected, tabulated, and statistically analysed using a Pair-wise comparisons test and the Kruskal-Wallis test. Maximum biting force was tested at baseline,3 months, 6 months, and 12 months for each group; the results were collected, tabulated, and statistically analysed using a Pair-wise comparisons test and ANOVA test.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with sufficient residual alveolar bone quantity and quality anterior to the mental foramen to receive self-taping root form titanium implants.
2. Maxillary and Mandibular residual alveolar ridges covered with healthy mucosa without any remaining roots or local inflammation.
3. Patients with sufficient inter-arch space (at least 15 mm) to have overdenture and bar attachment.
4. U-shaped lower ridge to avoid the lingual placement of the bar that occurs with a V-shaped ridge.
5. Patients with skeletal and dental class I.

Exclusion Criteria:

1. Patients with systemic diseases such as cardiovascular diseases, any disease of immunity, febrile conditions such as epilepsy, metabolic disorders, osteoporosis, hyperparathyroidism, and impaired psychological conditions that might affect the oral tissues or the bone metabolic rate.
2. Patients with local and general contraindications for surgical procedures.
3. Patients with TMJ or neuromuscular disorder.
4. Patients with Para functional habits such as bruxism and clenching.
5. Patients with impacted teeth or remaining roots.
6. Alcoholic patients.
7. Patients with a history of radiotherapy in the head and neck region.
8. Non-cooperative patients.
9. Patients with a history of bisphosphonate intake.
10. Patients with flabby tissues, bony undercuts, sharp bony edges, thin ridges or abnormalities at the lower alveolar ridge and recent extraction.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | 1 year
  questionnaire

SECONDARY OUTCOMES:
maximum biting force | 1 year
  occlusal force meter

CONTACTS AND LOCATIONS:
Overall Officials: Amr E Badr, phd, Study Chair — professor
Locations (1):
- Minia University, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
This randomised controlled clinical trial assessed patient satisfaction and maximum biting force with three differently constructed bar-retained overdentures (conventional casting, Milling and 3D printing CAD/CAM techniques) within a one-year follow-up.

REFERENCES:
- [Derived] Badr AMI, Nabawy M, Mohammed GF, Radwan SA. Evaluation of patient satisfaction and maximum biting force of three differently constructed bars on two implants retaining mandibular overdenture - one year follow-up (a randomized controlled clinical trial). BMC Oral Health. 2024 Nov 9;24(1):1360. doi: 10.1186/s12903-024-05092-x. PMID 39522003